CLINICAL TRIAL: NCT01160549
Title: Study of Pregnancy Hormone Concentrations in Urban and Nomadic Mongolian Women
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910152; 10-C-N152
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy
Keywords: Pregnancy; Hormones; Mongolia; Asian; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Women living in rural environments
- Controls: Women living in more urban environments

SUMMARY:
International variation in breast cancer rates and data from migrant and animal studies support the possibility that exposures early in development, including the in utero period, play a role in breast carcinogenesis. One of the most striking prenatal influences on breast cancer risk is whether the woman was born in a country with a low or high breast cancer incidence. This observation has led to interest in the degree to which in utero exposures vary by the maternal environment, and to the hypothesis that alterations in prenatal concentrations of steroid hormones, particularly estrogens, and other biologic parameters to which the fetus is exposed mediate differences in subsequent breast cancer risk.

There are striking differences in breast cancer incidence rates between Asian and North American and Western European populations, but variation within Asia is also wide. Incidence in Mongolia is one of the lowest in the world (6.6/100,000) while China, its neighbor to the south, has about three times this rate (18.7/100,000). Furthermore, rates appear higher in urban than in rural areas. Over the last decade and a half Mongolia has experienced profound economic changes resulting in mass migration from a nomadic or semi-nomadic existence to a more western lifestyle in the capital city of Ulaanbaatar. Together with the contrast in exposures between traditional and urban settings, migration presents the opportunity to study women as they acculturate to a more western lifestyle.

We propose collecting maternal and cord blood samples from pregnant Mongolian women and their offspring living in rural and urban areas to describe concentrations of several steroid hormones and growth factors. The purpose of the study is to assess whether the in utero environment differs in women living a traditional lifestyle compared with a more urban lifestyle, and by degree of western acculturation among those who have recently migrated to the capital. Maternal and cord blood samples from an ongoing cohort study being conducted at the University of Pittsburgh will provide a comparison group of US women.

DETAILED DESCRIPTION:
The National Cancer Institute has been conducting research in countries around the world with the purpose of documenting international differences in hormone and growth factor levels with the intent of trying to understand how these relate to health. In particular, recent evidence suggests that hormones and growth factors very early in life may affect later disease risk. Dr. Ganmaa, a native Mongolian physician and Harvard-trained scientist suggested including Mongolia as one of the research settings for the NCI multi-centered study since the country offers a distinct population with unique lifestyles and traditions.

Over the last decade and a half Mongolia has experienced profound economic changes resulting in mass migration from a nomadic or semi-nomadic existence to a more western lifestyle in the capital city of Ulaanbaatar. Together with the contrast in exposures between traditional and urban settings, migration presents the opportunity to study women as they acculturate to a more western lifestyle.

Mongolia provides a unique opportunity to assess whether differences in urban and rural lifestyles and behaviors influence health. The purpose of the study is to assess whether the pregnancy environment differs in women living a traditional lifestyle compared with a more urban lifestyle, and by degree of western acculturation among those who have recently migrated to the capital. We plan to compare steroid hormones and growth factors in maternal and cord blood samples from pregnant Mongolian women living in rural and urban areas with pregnant women from the US (at Brigham and Women's Hospital in Boston), UK (the Avon Longitudinal Study of Parents and Children), Norway (the Norwegian Mother and Child Cohort) and outside Beijing, China (CDC's randomized trial of pregnancy supplements).

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible for study are pregnant women 18 years of age or older, with singleton, presumed to be viable pregnancies that were naturally conceived, who receive prenatal care at the Maternity Hospital in UlaanBaatar (MCHRC) or the Bulgan and Selenge General Hospitals.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Maternal and cord blood samples from pregnant Mongolian women and their offspring living in rural and urban areas (by administrative divisions, called aimags).
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2015-02-19 (Actual)

PRIMARY OUTCOMES:
Hormone measurements | Cross sectionally
  Assess whether the in utero environment differed in women living a traditional lifestyle compared with a more urban lifestyle, and by degree of Western acculturation among those who had recently migrated to the capital. In addition, we planned to study the endocrine profile of pre-menopausal women living in UlaanBaatar by their migration status among mothers of girls participating in a study of milk consumption and hormonal status conducted by our collaborators at Harvard Medical School. Reproductive hormones were measured and are being compared to those in women living in the UK.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Troisi, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- Mongolia (4):
  - National University of Mongolia, School of Social Science, Baga Toirog
  - Bulgan General Hospital, Ulaanbaatar
  - Maternal and Child Health Research Center (MCHRC), Ulaanbaatar
  - Selenge General Hospital, Ulaanbaatar

REFERENCES:
- [Background] Ahsan H. Placental genes and breast cancer: can the offspring's or father's genotypes predict mother's risk? Epidemiology. 2003 Mar;14(2):251-3. doi: 10.1097/01.EDE.0000050696.19411.C0. PMID 12606894
- [Background] Atamer Y, Erden AC, Demir B, Kocyigit Y, Atamer A. The relationship between plasma levels of leptin and androgen in healthy and preeclamptic pregnant women. Acta Obstet Gynecol Scand. 2004 May;83(5):425-30. doi: 10.1111/j.0001-6349.2004.00276.x. PMID 15059152
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258